CLINICAL TRIAL: NCT04826250
Title: The Effect of Timing of Antihypertensive Medication on Diurnal Fluctuations in Blood Pressure Using a Wearable Sensor With Continuous Monitoring
Acronym: ABPM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary data was not sufficient to support the study aim
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Gepner Yftach, Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ABPM
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Hypertension
Keywords: ambulatory blood pressure monitoring; diurnal fluctuations; cardiovascular risk; Hypertension; wireless monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertensive patients - nighttime medication (Experimental): Hypertensive patients will be instructed to take their medication in the evening for four consecutive weeks. At the end of this period, participants will switch the timing of medication to the morning for four weeks.
  Interventions: Procedure: Timing of medication
- Hypertensive patients - morning medication (Experimental): Hypertensive patients will be instructed to take their medication in the morning for four consecutive weeks. At the end of this period, participants will switch the timing of medication to the evening for four weeks.
  Interventions: Procedure: Timing of medication

INTERVENTIONS:
Procedure: Timing of medication — Either morning or nighttime medication

SUMMARY:
Minimal or absent of diurnal fluctuation in blood pressure, and specifically conditions in which BP values are elevated during the night compared to daytime (rather than "nighttime dipping"), are associated with higher rates of morbidity and all-cause mortality. However, there is a gap in the scientific literature as to the optimal, individualized, timing of administration of antihypertensive drugs to balance daytime/nighttime fluctuations in BP to reduce the risk for cardiovascular morbidity and all-cause mortality.

To date, the most widely used method for semi-continuous, ambulatory monitoring of BP is a Holter, cuff-based monitor, which is cumbersome to use and therefore results in low patient compliance. Despite various attempts to overcome this problem, practical, patient-friendly methods for continuous BP monitoring throughout the day and night are currently not available.

Thus, the main of this study was to investigate whether there is a differential effect of timing of administration of antihypertensive drugs on diurnal fluctuations in BP using a wearable, cuff-less sensor with continuous monitoring capabilities. It is hypothesized that evening medication will improve BP fluctuations throughout the day (e.g., allow nighttime dipping and prevent morning surges) to a greater extend than morning meditation in people with hypertension.

DETAILED DESCRIPTION:
Elevated blood pressure (i.e., hypertension) is a major risk factor for cardiovascular morbidity and all-cause mortality. Medical treatment can significantly improve the prognosis of those with hypertension. It has also been suggested that nighttime medication is more effective in improving mortality and morbidity compared to daytime medication. This hypothesis relates to the fact that lack of a reduction in BP during the night (termed "non-dipping") is associated with a worse prognosis, and therefore nighttime medication can potentially improve the desired diurnal fluctuations in BP and improve health outcomes in those with hypertension to a greater extent than daytime medication. However, whether the timing of drug administration affects the desired diurnal fluctuations in BP remains unknown.

To assess fluctuations in BP throughout the day, and specifically during the night, an ambulatory BP monitoring (ABPM) for 24 hours is required. Research suggests that this method allows classification of hypertension and thus more precise prediction of the patient's cardiovascular risk compared to office-based BP monitoring.

To date, clinician's ability to continuously monitor BP throughout the day has been limited, as the mostly commonly used method of Holter monitoring only allows for BP measurement every 30 min and imposes a significant burden on the patient. The latter limitation affects patients' compliance, and thus clinicians' ability to accurately assess daily BP fluctuations (or lack thereof) that present a major health risk factor.

Thus, the main aim of this study is to use a new wearable, cuff-less technology that that allows continuous ambulatory monitoring of BP to assess whether nighttime medication for hypertension improved diurnal fluctuations in BP to a better extent compared to daytime medication.

Methods:

This is interventional, cross-over and randomized study will be performed in a medical hospital. One hundred and fifty hypertensive patients, ages 30-80, will be recruited by a practicing medical physician and perform baseline tests that include blood work and BP measurement, as well as 24 monitoring of physiological signs (e.g., heart rate, BP, cardiac output and index and vascular resistance) using a photoplethysmogram (PPG)-based wireless, wearable device to obtain baseline measures. Participants will then begin medical treatment, either in the morning or evening, for four weeks. Physiological signs will again be continuously monitored using the wireless device during the last 48 hours of this time-period. After four weeks, participants will switch the timing of their medication for four more week, including 48 hours of monitoring.

Blood pressure measurement: BP will be continuously collected using a wearable, non-invasive, wireless chest-monitor (Biobeat Technologies Ltd., Petah Tikva, Israel), that is based on PPG technology. Systolic and diastolic BPs will be monitored and recorded continuously for the last 48 hours of each four-week intervention and compared between morning and evening medication, for each participant (i.e., each participant will serve as their own control).

Blood tests: Blood work will be performed after a 12-hour fast at baseline and at the end of each intervention. Measured parameters such as glucose, insulin, low and high density lipoprotein cholesterol, total cholesterol ,triglycerides sodium and potassium will enable assessment of cardio-metabolic risk.

Questionnaires: life quality and sleep quality questionnaires will be administered at baseline and at the end of each intervention

ELIGIBILITY:
Inclusion Criteria:

* Hypertension

Exclusion Criteria:

* hypertensive emergency
* Those taking more than 3 anti-hypertensive drugs
* congestive heart failure
* pregnancy
* renal failure

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Nighttime blood pressure | Baseline
  blood pressure measured during the night
Nighttime blood pressure | At the end of the first four-week intervention
  blood pressure measured during the night
Nighttime blood pressure | At the end of the second four-week intervention
  blood pressure measured during the night
morning blood pressure | Baseline
  blood pressure measured during the morning hours
morning blood pressure | At the end of the first four-week intervention
  blood pressure measured during the morning hours
morning blood pressure | At the end of the second four-week intervention
  blood pressure measured during the morning hours

SECONDARY OUTCOMES:
Blood Glucose | Baseline
  Blood parameters indicative of cardio-metabolic health
Blood Glucose | At the end of the first four-week intervention
  Blood parameters indicative of cardio-metabolic health
Blood Glucose | At the end of the second four-week intervention
  Blood parameters indicative of cardio-metabolic health
Insulin | Baseline
  Blood parameters indicative of cardio-metabolic health
Insulin | At the end of the first four-week intervention
  Blood parameters indicative of cardio-metabolic health
Insulin | At the end of the second four-week intervention
  Blood parameters indicative of cardio-metabolic health
Low and high density lipoprotein cholesterol, total cholesterol, triglycerides | Baseline
  Blood parameters indicative of cardio-metabolic health
Low and high density lipoprotein cholesterol, total cholesterol, triglycerides | At the end of the first four-week intervention
  Blood parameters indicative of cardio-metabolic health
Low and high density lipoprotein cholesterol, total cholesterol, triglycerides | At the end of the second four-week intervention
  Blood parameters indicative of cardio-metabolic health
Sodium, potassium | Baseline
  Blood parameters indicative of cardio-metabolic health
Sodium, potassium | At the end of the first four-week intervention
  Blood parameters indicative of cardio-metabolic health
Sodium, potassium | At the end of the second four-week intervention
  Blood parameters indicative of cardio-metabolic health

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel